CLINICAL TRIAL: NCT00831896
Title: A Multicenter, Open-Label, Dose Escalation Phase I Study of TAK-701 in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: Phase I Study of TAK-701 in Adult Patients With Advanced Nonhematological Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C17001
Record Dates: First submitted 2009-01-26; First posted 2009-01-29 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2011-12

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): TAK-701
  Interventions: Biological: TAK-701

INTERVENTIONS:
Biological: TAK-701 — Either 2, 5, 10, or 20 mg/kg IV. Cycle 1: single dose at 2x the dose assignment; Cycle 2 and beyond: dose once every two weeks
  Dosing continues until disease progression, unacceptable toxicity related to TAK-701, or maximum of 12 cycles, unless determined that patient would benefit from continued therapy.

SUMMARY:
This study is a multicenter, open-label, dose escalation, phase 1 study of TAK 701 in adult patients with advanced nonhematologic malignancies. This study will be the first to administer TAK 701 to humans. The primary purpose of this study is to determine the safety profile, tolerability, and pharmacokinetics profile of TAK-701.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 years or older.
2. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
3. Diagnosis of a nonhematologic malignancy for which standard curative or lifeprolonging treatment does not exist or is no longer effective.
4. Radiographically or clinically evaluable tumor; however, measurable disease is not required for participation in this study (eg, patients with pleural effusion or ascites).
5. Female patients who:

   * Are postmenopausal for at least 1 year before the screening visit, or
   * Are surgically sterile, or
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent form through 3 months after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.

   Male patients, even if surgically sterilized (ie, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study drug treatment period and through 3 months after the last dose of TAK-701, or
   * Agree to completely abstain from heterosexual intercourse.
6. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

1. Female patients who are lactating or have a positive serum pregnancy test during the screening period.
2. Major surgery within 14 days before the first dose of TAK-701 or any planned/anticipated surgery during the study period.
3. Positive test for Hepatitis B or C infection.
4. Active alcohol abuse
5. Active infection requiring systemic therapy, or other serious infection.
6. Antineoplastic therapy (including unconjugated therapeutic antibodies and toxin immunoconjugates) or any experimental therapy within 21 days before the first dose of TAK-701.
7. Radiotherapy within 21 days before the first dose of TAK-701.
8. Nitrosoureas or mitomycin-C within 6 weeks before the first dose of TAK-701.
9. Autologous stem cell transplant within 3 months before the first dose of TAK-701, or prior allogeneic stem cell transplant at any time.
10. Any prior exposure to anti-HGF therapy (eg, AMG-102, AV-299).
11. The patient has symptomatic brain metastasis.
12. Absolute neutrophil count < 1,500/mm3; platelet count < 100,000/mm3.
13. Calculated creatinine clearance < 50mL/minute
14. Any of the following clinical laboratory results during screening (ie, within 28 days before the first dose of TAK-701):

    * Bilirubin > 1.5 times the upper limit of the normal range (ULN).
    * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 times the ULN. AST and ALT may be elevated up to 5 times the ULN if their elevation can be reasonably ascribed to the presence of metastatic disease to liver and/or to bone.
15. Known human immunodeficiency virus (HIV) positive.
16. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
17. Uncontrolled cardiovascular condition, including ongoing cardiac arrhythmias, congestive heart failure, angina, or myocardial infarction within the past 6 months.
18. Patients having QTc > 470 msec on a 12-lead ECG obtained within 28 days before first study drug administration.
19. Presence of serious or nonhealing wound, ulcer or bone fracture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-03; Primary Completion 2010-11 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety profile (adverse events including dose limiting toxicities, clinical safety assessments such as human antihumanized antibody (HAHA) and neutr. HAHA), tolerability (maximum tolerated dose or maximum feasible dose), and pharmacokinetic profile. | Duration of study

SECONDARY OUTCOMES:
Pharmacodynamic profile, cardiac repolarization effects, antitumor activity, and recommended Phase 2 dose of TAK-701 | Duration of study
Investigator's assessment of disease response using Response Evaluation Criteria in Solid Tumors guidelines and relevant tumor markers in serum such as PSA, CA 125 and CA 19-9 | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (3):
- United States (3):
  - Emory University School of Medicine, Winship Cancer Institute, Atlanta, Georgia
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The Sarah Cannon Research Institute, Nashville, Tennessee